CLINICAL TRIAL: NCT02260453
Title: Randomized Controlled Trial Analyzing the Role of Systematic Preoperative Coronary Angiography Before Elective Carotid Endarterectomy in Patients With Asymptomatic Coronary Artery Disease
Brief Title: Coronary Angiography Before Elective Carotid Endarterectomy in Patients With Asymptomatic Coronary Artery Disease
Acronym: CACEA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Giulio Illuminati, Associate Professor of Surgery, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: University "La Sapienza" Rome
Record Dates: First submitted 2014-10-06; First posted 2014-10-09 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Carotid Stenosis; Coronary Stenosis
MeSH Terms: conditions — Carotid Stenosis; Coronary Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A - Coronary angiography (Active Comparator): All the patients receive preoperative coronary angiography followed, if needed, by percutaneous intervention (PCI) or bypass (CABG)
  Interventions: Other: Preoperative coronary angiography
- B - standard cardiac workup (Active Comparator): Standard cardiac workup
  Interventions: Other: Standard cardiac workup

INTERVENTIONS:
Other: Preoperative coronary angiography — If coronary disease is detected percutaneous intervention (PCI) or coronary artery bypass grafting (CABG) is applied
  Arms: A - Coronary angiography
Other: Standard cardiac workup — EKG, transthoracic cardiac echocardiogram
  Arms: B - standard cardiac workup

SUMMARY:
The purpose of this study is to evaluate the potential benefit of systematic preoperative coronary angiography followed by selective coronary artery revascularization on the incidence of myocardial infarction (MI) in patients without a history of coronary artery disease (CAD) and undergoing carotid endarterectomy (CEA).

DETAILED DESCRIPTION:
Patients candidates for CEA, with no history of CAD, a normal electrocardiogram (ECG), and a normal cardiac ultrasound were randomized in two groups. In group A (n = 216) all patients underwent coronary angiography before CEA +- coronary artery revascularization. In group B (n = 210) CEA was performed without coronary angiography.

ELIGIBILITY:
Inclusion Criteria:

* indication for carotid endarterectomy
* no clinical sign or history of ischemic heart disease
* no electrical signs of cardiac ischemia
* left ventricular ejection fraction >50% at transthoracic echocardiogram.

Exclusion Criteria:

* disabling stroke (mRS ≥3)
* non atherosclerotic carotid disease
* severe intracranial carotid artery stenosis
* contra-indications to heparin, aspirin or clopidogrel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 426 (Actual)
Dates: Start 2005-01; Primary Completion 2009-07 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Non-fatal and fatal myocardial infarction | 30 days through year 3

SECONDARY OUTCOMES:
All-cause and cardiovascular mortality | 30 days through year 3

CONTACTS AND LOCATIONS:
Overall Officials: Giulio Illuminati, MD, Principal Investigator — University of Roma La Sapienza

REFERENCES:
- [Derived] Illuminati G, Schneider F, Greco C, Mangieri E, Schiariti M, Tanzilli G, Barilla F, Paravati V, Pizzardi G, Calio' F, Miraldi F, Macrina F, Totaro M, Greco E, Mazzesi G, Tritapepe L, Toscano M, Vietri F, Meyer N, Ricco JB. Long-term results of a randomized controlled trial analyzing the role of systematic pre-operative coronary angiography before elective carotid endarterectomy in patients with asymptomatic coronary artery disease. Eur J Vasc Endovasc Surg. 2015 Apr;49(4):366-74. doi: 10.1016/j.ejvs.2014.12.030. Epub 2015 Feb 18. PMID 25701070